CLINICAL TRIAL: NCT06338085
Title: The Effect of Emotional Freedom Technique on Depressive and Menopausal Symptoms in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meryem Vural Şahin (Other)
Responsible Party: Sponsor-Investigator, Meryem Vural Şahin, Phd Student, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: meryemvrlshn00000000002
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Menopause

STUDY DESIGN:
Intervention Model Description: the groups with a conventional therapy control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The researcher will provide the intervention group with Emotional Freedom Technique (EFT) training, which will last for 2 sessions of 45 minutes with 1 day intervals.Participants will then be asked to continue the techniques taught during the training on their own once a day for 8 weeks.
  Interventions: Other: emotional liberation technique
- control group (No Intervention): no intervention will be made to the control group

INTERVENTIONS:
Other: emotional liberation technique — In this intervention, with the technique taught by the researcher, women will self-administer the practice of lightly touching certain points 5 days and 1 time per week for 8 weeks. A whatsup group will be created by the researcher. A reminder message will be sent from this group to do the practice 1 time every day.
  Arms: intervention group

SUMMARY:
The aim of this study is to determine the effect of EFT (Emotional Freedom Technique), a nonpharmacological method, on menopausal symptoms and depression in postmenopausal women. By determining the effectiveness of the Emotional Freedom Technique, the applicability of non-pharmacological method treatment in women with depression and menopausal symptoms in postmenopausal period will be proven. As a result of the study, if a positive effect on menopausal symptoms and depression is found in women with EFT, it can be recommended as an evidence-based alternative method in midwifery and nursing care.

DETAILED DESCRIPTION:
Menopausal period is defined as the stage of transition to old age, which starts with the decline in ovarian function and decrease in reproductive capacity and ends with the end of reproductive ability over time. According to the WHO definition, natural menopause is the permanent cessation of menstruation with the loss of ovarian activity. The average age of menopause worldwide is 51 years and the transition to menopause occurs between the ages of 45 and 55. Menopause is defined after a 12-month amonereal period. Induced menopause is the cessation of menstruation as a result of surgical removal of both ovaries or external factors such as chemotherapy and radiotherapy. Before the age of 40, cessation of menstruation is defined as early menopause.

Approximately one-third of women experience no or mild symptoms during menopausal life, one-third experience moderate symptoms, and the remaining one-third may experience severe symptoms.The symptomatology experienced during this period is characterized by a hypoestrogenic state that occurs due to the decline in ovarian function in 60% to 80% of women. With menopause; estradiol level decreases 5-10 times, testosterone level decreases, follicle stimulating hormone (FSH) level increases 10-20 times and luteinizing hormone (LH) increases 3 times. As a result of insufficient secretion of sex hormones in women during this period, insomnia, vaginal dryness, irregular menstruation, depressive mood, irritability, headache, forgetfulness, dizziness, and vasomotor symptoms such as changes in body thermoregulation and night sweats may be observed. The experience of menopausal symptoms is individual and depends not only on hormonal changes but also on external factors such as living conditions, general health, social functioning and perceptions of aging. These factors can influence the perception and assessment of menopause.

The menopausal period is associated with various biopsychosocial changes, and some women may have physical and psychological symptoms of different severity. Increasing evidence suggests that increased sensitivity to estradiol fluctuation plays an important role in the development of depressive symptoms during the menopausal transition. A meta-analysis of 11 studies found that perimenopause is a period in which women are more likely to experience depressive symptoms compared to other menopause periods. In a descriptive study conducted to determine the quality of life in 99 perimenopausal women aged 45-55 years, almost all women experienced physical and psychosocial symptoms, while severe vasomotor symptoms and psychosocial symptoms were found in women who could not manage stress.

Depression affects approximately 350 million people worldwide and is a global burden. Depression is twice as common in women compared to men and the risk of depression may increase during periods of hormonal changes such as puberty, pregnancy and menopause. Although it is not specifically stated that there is a definite relationship between hormonal changes and depression, hormonal changes in the stages of women's life are called risky periods. Although the menopausal period, when hormonal changes are intense, is not associated with psychiatric disorders alone, it may increase the risk of a history of depressive disorder, especially in women in the perimenopausal period. Absolute levels and fluctuations of hypothalamic-pituitary-gonadal hormones during menopause are possible predictors of mood disorders and depression in perimenopause.

In a cross-sectional study conducted in Switzerland with 114 women aged 40-56 years, menopausal symptoms were significantly associated with perimenopausal depressive symptoms. As a result of a study on Women's Health Needs in China, in which 3199 women aged 40-55 years were examined, the prevalence of depressive symptoms was 19.3%, while there was a significant relationship between menopausal symptoms and depressive symptoms. In a descriptive study conducted with 176 women aged 45 to 60 years in Korea, it was determined that menopausal symptoms significantly affected depression status. In a descriptive study conducted with 749 women aged 45-60 years in Brazil, it was determined that moderate menopausal symptoms were significantly associated with depression or anxiety. Elaslan (2018) found that 64.4% of menopausal women aged 45-55 years experienced physical-psychological problems. Aygün (2019) conducted a study with 112 women aged 40-64 years and found that 25% of women had depression, while those who entered menopause had higher depression scores than those who did not.

and emotional liberation techniques in the treatment of depression. Emotional Freedom Technique (EFT) is a brief and evidence-based intervention that combines elements of acupressure point exposure, cognitive therapy and somatic stimulation on the face and body. Participants' distress about any issue or situation is determined. They are asked to rate their level of distress on a Likert-type scale out of 10 (10 representing maximum distress and 0 representing minimum distress). This is called the Subjective Distress Unit (SUDS) scale. Participants then indicate their concerns in a 'Set-up Statement' which helps to translate them into their own level of distress. This is usually expressed as: "Although I have this problem (e.g. anger), I accept myself deeply and completely." The first half of the Set-up Statement emphasizes the exposure, while the second half frames the traumatizing event in the context of self-acceptance. The participant then engages in somatic tapping on acupuncture points on the body while repeating an abbreviated phrase to stay engaged (e.g., feeling angry). This is called the "Reminder Phrase". The tapping sequence uses 8 acupoints on the face and upper body and is normally repeated until the SUDS rating is very low (1 or 0). In order for the EFT treatment outcome to be successful, the method is usually performed between four and 10 sessions. Comorbid conditions such as anxiety and depression improve simultaneously. Contributes to the regulation of biological markers such as stress hormones. The risk of adverse events is low. The application provides psychological as well as physiological improvements. The method can be used in online and telemedicine applications.

Emotional Freedom Technique (EFT) is defined as a clinical procedure that nurses can offer to patients to relieve psychological and physical distress. EFT is a therapy that combines cognitive and somatic elements. It can effectively treat physiological and psychological symptoms. This therapy helps the person to calm down after lightly tapping on certain points. As a result of the systematic review study conducted to determine the effect of EFT, the Emotional Freedom Technique for Pain, Anxiety Disorders and Depression, it was determined that it is a therapy that can affect physiological symptoms, pain, anxiety disorders and depression. It is recommended to apply EFT as a method of clearing the mind, focusing (such as meditation) and improving attitudes to better cope with emotional problems. In a study conducted to determine the effect of EFT on menopausal symptoms in women with breast cancer receiving hormonal treatment, women (n=41) were given EFT training for 3 hours a week for 3 weeks. Then, they practiced EFT on themselves for 9 weeks. At the end of the study, a significant decrease in the degree and number of hot flashes among menopausal symptoms and a significant decrease in anxiety and depression scores were found. In a study conducted to determine the effect of EFT on depression in patients diagnosed with depression, 100 participants were divided into two separate groups. The intervention group received 40 minutes of EFT for three consecutive days in addition to routine treatment. The other group received only conventional treatment. As a result of the study, the depression scale score of the intervention group decreased more than before the treatment. The effect of EFT on depression According to the results of the meta-analysis study in which 20 studies were included, it was determined that EFT treatment given individually or as a group for depression was superior to psychopharmacology and psychotherapy. As a result of the meta-analysis study conducted to examine the effectiveness of EFT application used in the treatment of post-traumatic stress disorder (PTSD), it was determined that the effect size of EFT application on PTSD, anxiety and depression was significant. In the RCT examining the effect of EFT on postmenopausal depression in menopausal women, 88 women with mild and moderate depression were divided into two groups. Those in the intervention group received 2 sessions of EFT training. Then, they were asked to continue EFT practice once a day for 8 weeks. The control group received training on sham acupressure points. As a result of the study, it was determined that 8-week EFT practice significantly reduced depression scores in postmenopausal women.

The menopausal period is one of the most challenging and important phases of a woman's life. This period can be a troublesome time when women may experience physical and psychological changes and some problems. Women's physical and psychosocial health can be negatively affected. This negative situation can affect not only the woman but also the family and society. According to Tuik 2019 data, life expectancy in women was determined as 81.3 years. Considering the life expectancy in women, women spend a significant part of their lives in the menopausal period. Therefore, it is important to treat menopausal and depressive symptoms experienced during this period. In the menopausal period, not only medical treatment is not sufficient, but effective and qualified counseling and non-pharmacological methods are used.

ELIGIBILITY:
Inclusion Criteria:

* Being in menopausal period (no menstruation in the last 12 months)
* Literacy,
* No visual, auditory and mental disabilities

Exclusion Criteria:

* Receiving cancer treatment during research,
* Diagnosed with depression during the research,
* Taking any psychiatric medication during the study,
* Receiving hormone replacement therapy before or during the trial
* Who did not attend the Eft sessions

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Scale | 8 weeks
  It was developed in 1961 by Beck et al. Reliability and validity analysis in Turkey was conducted by Hisli et al. in 1988. The scale consists of 21 questions. Each question is scored between 0-3 points. The total score that can be obtained from the scale is between 0-63. A high score on the scale increases the severity of depression. A score between 10-17 points indicates mild depression, 18-29 points indicates moderate depression, and a score between 30-63 points indicates severe depression. In the Turkish validity analysis of the scale, Cronbach's alpha coefficient was found to be 0.74.

SECONDARY OUTCOMES:
Menopause Rating Scale (MRS) | 8 weeks
  Menopause Rating Scale (MRS) was developed by Schneider et al. to measure the severity of menopausal symptoms. It was adapted into Turkish by Gürkan in 2005. In the Likert-type scale consisting of a total of 11 items including menopausal complaints, there are "0= None", "1= Mild", "2= Moderate", "3= Severe" and "4= Very severe" options for each item. The total score of the scale is calculated based on the scores given for each item. The lowest score is 0 and the highest score is 44. An increase in the total score indicates an increase in the severity of the complaints. The Cronbach Alpha coefficient for the whole scale is 0.84.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem UĞURLU, Study Director — Gulhane School of Medicine
Locations (1):
- family health center no. 1 in Çayyolu, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambikairajah A, Walsh E, Tabatabaei-Jafari H, Cherbuin N. Fat mass changes during menopause: a metaanalysis. Am J Obstet Gynecol. 2019 Nov;221(5):393-409.e50. doi: 10.1016/j.ajog.2019.04.023. Epub 2019 Apr 26. PMID 31034807
- [Background] Ambikairajah A, Walsh E, Cherbuin N. A review of menopause nomenclature. Reprod Health. 2022 Jan 31;19(1):29. doi: 10.1186/s12978-022-01336-7. PMID 35101087
- [Background] Bustami M, Matalka KZ, Elyyan Y, Hussein N, Hussein N, Abu Safieh N, Thekrallah F, Mallah E, Abu-Qatouseh L, Arafat T. Age of Natural Menopause Among Jordanian Women and Factors Related to Premature and Early Menopause. Risk Manag Healthc Policy. 2021 Jan 19;14:199-207. doi: 10.2147/RMHP.S289851. eCollection 2021. PMID 33500673
- [Background] Curta JC, Weissheimer AM. Perceptions and feelings about physical changes in climacteric women. Rev Gaucha Enferm. 2020;41(spe):e20190198. doi: 10.1590/1983-1447.2020.20190198. Epub 2020 May 8. English, Portuguese. PMID 32401861
- [Background] Trimarco V, Rozza F, Izzo R, De Leo V, Cappelli V, Riccardi C, Di Carlo C. Effects of a new combination of nutraceuticals on postmenopausal symptoms and metabolic profile: a crossover, randomized, double-blind trial. Int J Womens Health. 2016 Oct 11;8:581-587. doi: 10.2147/IJWH.S115948. eCollection 2016. PMID 27785106
- [Background] Weidner K, Bittner A, Beutel M, Goeckenjan M, Brahler E, Garthus-Niegel S. The role of stress and self-efficacy in somatic and psychological symptoms during the climacteric period - Is there a specific association? Maturitas. 2020 Jun;136:1-6. doi: 10.1016/j.maturitas.2020.03.004. Epub 2020 Mar 13. PMID 32386660
- [Background] Li X, Ren Z, Ji T, Shi H, Zhao H, He M, Fan X, Guo X, Zha S, Qiao S, Li Y, Pu Y, Liu H, Zhang X. Associations of sleep quality, anxiety symptoms and social support with subjective well-being among Chinese perimenopausal women. J Affect Disord. 2022 Apr 1;302:66-73. doi: 10.1016/j.jad.2022.01.089. Epub 2022 Jan 24. PMID 35085670
- [Background] Mathew DJ, Kumar S, Jain PK, Shukla SK, Ali N, Singh DR. A Cross-Sectional Study to Assess the Quality of Life of Perimenopausal and Post menopausal Women in Rural Etawah, Uttar Pradesh, India. J Midlife Health. 2020 Jul-Sep;11(3):161-167. doi: 10.4103/jmh.JMH_88_19. Epub 2020 Sep 29. PMID 33384540
- [Background] Aygün, M. S.,(2019). Evaluation of the frequency and relationship between menopause and depression symptoms in women aged 40-64 years who applied to Ankara University family medicine outpatient clinics.
- [Background] Bach D, Groesbeck G, Stapleton P, Sims R, Blickheuser K, Church D. Clinical EFT (Emotional Freedom Techniques) Improves Multiple Physiological Markers of Health. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X18823691. doi: 10.1177/2515690X18823691. PMID 30777453
- [Background] Gordon JL, Halleran M, Beshai S, Eisenlohr-Moul TA, Frederick J, Campbell TS. Endocrine and psychosocial moderators of mindfulness-based stress reduction for the prevention of perimenopausal depressive symptoms: A randomized controlled trial. Psychoneuroendocrinology. 2021 Aug;130:105277. doi: 10.1016/j.psyneuen.2021.105277. Epub 2021 May 19. PMID 34058560
- [Background] Soares CN. Depression in peri- and postmenopausal women: prevalence, pathophysiology and pharmacological management. Drugs Aging. 2013 Sep;30(9):677-85. doi: 10.1007/s40266-013-0100-1. PMID 23801148
- [Background] Elsan, T. (2018). Evaluation of the quality of life of menopausal women applying to a PHC area (Master's thesis, Institute of Health Sciences).
- [Background] Deecher D, Andree TH, Sloan D, Schechter LE. From menarche to menopause: exploring the underlying biology of depression in women experiencing hormonal changes. Psychoneuroendocrinology. 2008 Jan;33(1):3-17. doi: 10.1016/j.psyneuen.2007.10.006. Epub 2007 Dec 3. PMID 18063486
- [Background] Baker, B. S., & Hoffman, C. J. (2015). Emotional Freedom Techniques (EFT) to reduce the side effects associated with tamoxifen and aromatase inhibitor use in women with breast cancer: A service evaluation. European Journal of Integrative Medicine, 7(2), 136-142.
- [Background] Willi J, Suss H, Grub J, Ehlert U. Biopsychosocial predictors of depressive symptoms in the perimenopause-findings from the Swiss Perimenopause Study. Menopause. 2021 Jan 4;28(3):247-254. doi: 10.1097/GME.0000000000001704. PMID 33399325
- [Background] Vivian-Taylor J, Hickey M. Menopause and depression: is there a link? Maturitas. 2014 Oct;79(2):142-6. doi: 10.1016/j.maturitas.2014.05.014. Epub 2014 Jun 2. PMID 24951102
- [Background] Augoulea A, Moros M, Lykeridou A, Kaparos G, Lyberi R, Panoulis K. Psychosomatic and vasomotor symptom changes during transition to menopause. Prz Menopauzalny. 2019 Jun;18(2):110-115. doi: 10.5114/pm.2019.86835. Epub 2019 Jun 28. PMID 31485208
- [Background] Church D, Stapleton P, Sabot D. App-Based Delivery of Clinical Emotional Freedom Techniques: Cross-Sectional Study of App User Self-Ratings. JMIR Mhealth Uhealth. 2020 Oct 14;8(10):e18545. doi: 10.2196/18545. PMID 32862128
- [Background] Mehdipour A, Abedi P, Ansari S, Dastoorpoor M. The effectiveness of emotional freedom techniques (EFT) on depression of postmenopausal women: a randomized controlled trial. J Complement Integr Med. 2021 May 19;19(3):737-742. doi: 10.1515/jcim-2020-0245. eCollection 2022 Sep 1. PMID 34013673